CLINICAL TRIAL: NCT06959472
Title: The Impact of Hyperarch Fascia Training on Ankle Sprain Pain and Exercise Performance in Athletic Men and Women
Brief Title: Impact of Hyperarch Fascia Training on Ankle Health and Exercise Performance
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Applied Science & Performance Institute (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: H030725
Record Dates: First submitted 2025-04-28; First posted 2025-05-06 (Actual); Last update posted 2025-06-03 (Actual); Status verified 2025-05

CONDITIONS: Ankle Injuries; Sprains and Strains; Joint Instability
Keywords: ankle sprain; ankle injury; ankle pain; ankle instability; remote rehabilitation; countermovement jump
MeSH Terms: conditions — Ankle Injuries; Sprains and Strains; Joint Instability

STUDY DESIGN:
Intervention Model Description: One group receives the Hyperarch Fascia Training (HFT) intervention.
  The other group (control) continues their regular activity without the HFT program.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hyperarch Fascia Training (HFT) Intervention Group (Experimental): Participants in this group will undergo a 12-week Hyperarch Fascia Training (HFT) program targeting foot and ankle fascial health. The protocol includes one weekly live 1-hour virtual session with a certified HFT coach and two independent 1-hour training sessions.
  Interventions: Behavioral: Hyperarch Fascia Training
- Control Group - Activities of Daily Living (ADL) (No Intervention): Participants in the control group will be instructed to maintain their usual activities of daily living (ADL) over the 12-week study period. They will not engage in any structured intervention or new rehabilitation protocol.

INTERVENTIONS:
Behavioral: Hyperarch Fascia Training — A 12-week behavioral intervention involving Hyperarch Fascia Training (HFT), which includes one weekly 1-hour virtual session with a certified coach and two 1-hour independent training sessions. The protocol combines meditation, mental imagery, foot and toe strengthening exercises, myofascial rolling, balance drills, and low-impact plyometrics.
  Arms: Hyperarch Fascia Training (HFT) Intervention Group

SUMMARY:
The purpose of this clinical trial is to evaluate whether the Hyperarch Fascia Training (HFT) program can reduce ankle pain and improve jump performance in active adults aged 20-45 with a history of ankle sprains. Participants will be randomly assigned to either an HFT intervention group or a control group, maintaining regular activity. Over 12 weeks, participants will complete remote training sessions, track jump performance using the "My Jump Lab" app, and complete ankle pain and stability questionnaires. All activities and assessments will be conducted remotely with guidance from certified coaches.

DETAILED DESCRIPTION:
This is a decentralized, randomized controlled trial evaluating the effects of Hyperarch Fascia Training (HFT) on pain and functional outcomes in adults aged 20-45 with a history of chronic ankle sprains. Up to 62 participants will be remotely recruited across the United States, with a target of 50 completing the study. Participants will be randomized to either an HFT intervention group or a passive control group, maintaining usual activity. The HFT group will complete three training sessions per week (one live virtual session and two self-guided sessions) over a 12-week period. Outcomes will assess pain and self-reported functional improvement using validated questionnaires and remote performance measures. All study activities, including recruitment, training, and assessments, will be conducted virtually.

ELIGIBILITY:
Inclusion Criteria:

* Gender: Male or females
* Age: 20-45 years old
* History of Chronic Ankle Sprains has led to present symptoms such as current pain and/or instability during weight-bearing activities, but no reported chronic knee, hip, or groin issues (within the past 3-months).
* Cumberland Ankle Instability Tool (CAIT) score ≤ 25, indicating significant instability in at least one ankle (Wright et al. 2014).
* Participants will be either recreationally trained, or considered trained/developmental as defined by McKay et al. (2021). Specifically, recreationally trained will be defined as meeting the World Health Organization (WHO) minimum activity guidelines of: minimal activity of at least 150-300 minutes of moderate-intensity activity, or 75-150min of vigorous-intensity activity a week; plus, muscle-strengthening activities 2 or more days a week. Recreationally trained participants may also participate in multiple sports/forms of activity. Trained/developmental will be defined as regularly training ~3 times per week, identifying with a specific sport, training with a purpose to compete. There is no performance standard required for these tiers.
* Health Status: Free from chronic diseases, cardiovascular conditions, and musculoskeletal injuries unrelated to ankle sprains.
* Be willing to attend a weekly one hour virtual training session on HFT plus a written program to be performed individually in two sessions for an additional 2 hours per week performed on their own. In total, be willing to train for up to 3-5 hours weekly on ankle rehabilitation.
* Agree to maintain their usual activity levels and avoid additional treatment modalities for the duration of the study.
* Have a iPhone smart phone XR (2018), or later model
* Have a desktop computer or laptop, with a camera for video conference calls and online training.
* Have a location with a minimum of 10ft * 10ft space for exercise movement, and appropriate ceiling height for vertical jump testing.

Exclusion Criteria:

* History of Achilles tendon rupture or surgery within the last 12 months. Use of prescribed corticosteroids or other tendon-specific treatments within four weeks prior to the study.
* Current enrollment in any structured fascial or tendon rehabilitation programs.
* Pregnancy, breastfeeding, or plans to become pregnant during the study period.
* Any medical conditions that may interfere with running or exercise performance or study participation.
* Not willing to sign an NDA regarding the fascia training techniques used in this study
* Use of medical interventions, such as growth hormone or peptides, that may influence tissue adaptation to exercise.
* Current supplementation with common soft-tissue ingredients, such as glucosamine, chondroitin, methylsufonylmethane (MSM), or collagen protein.
* Presents with Ehlers-Danlos syndrome (EDS) or hypermobility History or current drug abuse
* History or current cigarette smoke (including vaping) within the past 14 days from the screening visit
* Insulin-dependent diabetes and/or metformin use
* Chronic kidney or liver disease
* Has significant concurrent illnesses (controlled or uncontrolled), such as diabetes, lupus, epilepsy, or cardiac disorders, hepatitis B/C, HIV, serious mental health illness such as dementia or schizophrenia; psychiatric hospitalization in the past two years, or other, which in the opinion of the investigator, such conditions might be aggravated as a result of treatment
* Clinically diagnosed as depressed or taking depression or anti anxiety medication
* The investigator feels that for any reason the subject is not eligible to participate in the study
* History of uncontrolled cardiovascular disease (i.e., myocardial infarction, hypertension, hypercholesterolemia, peripheral vascular disease, other)
* Developmental disability or cognitive impairment that would preclude adequate comprehension of the informed consent form and/or ability to follow study subject requirement and/or record the necessary study measurements
* Currently has been diagnosed with cancer or has been in remission for less than 1 year
* Participation in any other investigational study within 30 days prior to consent.

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 62 (Estimated)
Dates: Start 2025-05-07 (Actual); Primary Completion 2025-10 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
Change in Aggregate Score on Cumberland Ankle Instability Tool (CAIT) | Baseline (Week 0), Week 8, and Week 12
  The CAIT is a 9-item self-reported questionnaire used to measure perceived ankle instability. Scores range from 0-30, with lower scores indicating greater instability.
Change in Aggregate Score on Foot and Ankle Ability Measure (FAAM) | Baseline (Week 0), Week 8, and Week 12
  The FAAM assesses functional ability with two subscales: Activities of Daily Living (ADL) and Sports. Each item is scored from 0 (unable to perform) to 4 (no difficulty), with higher scores indicating better function.

SECONDARY OUTCOMES:
Change in Countermovement Jump (CMJ) Performance | Baseline (Week 0), Week 8, and Week 12
  The performance measures for CMJ will include: Jump height, flight time, force, velocity, and power. Testing will begin with a standardized warm-up consisting of two sets of 10 bodyweight squats, with ~30 seconds of rest between each set. After warming up, participants will perform two maximal CMJs at their perceived maximal effort, with the highest performance being used as the outcome score. Data collection will involve recording all jumps using a mobile phone camera mounted on a tripod to capture motion in the frontal plane. The recordings will utilize artificial intelligence algorithms for markerless motion tracking at 60 Hz with a resolution of 1080p, processed through the previously validated "My Jump Lab" mobile application. To register CMJ performance, participants will be instructed to place their hands on their hips, look directly at the camera, and remain steady until the recording begins and then perform a maximal CMJ.
Change in Aggregate Score on Short Form Health Survey (SF-12) | Baseline (Week 0), Week 8, and Week 12
  The SF-12 measures quality of life across physical and mental health domains. Higher scores indicate better well-being .Question responses range from 1 to 5 or from 1 to 6 and each response is converted to a score from 0 to 100. For all questions, higher scores demonstrated greater well-being.
Glute Activation via Elevated Towel Curls | Baseline (Week 0), Week 8, and Week 12
  Participants will self-assess glute activation following the performance of elevated towel curls. At the end of this exercise, subjects rate below on a scale of 1-10 how much they feel this exercise activates (causes muscular tension) in their glutes. With 1 being no glute activation (no glute muscle tension) and 10 being complete glute activation (extreme glute muscle tension).

OTHER OUTCOMES:
Frequency and Nature of Adverse Events | Continuous throughout the 12-week intervention
  Self-reported or observed adverse events will be recorded and assessed for severity, causality, and frequency across both groups.

CONTACTS AND LOCATIONS:
Overall Officials: Jacob Wilson, PhD, Principal Investigator — Applied Science & Performance Institute
Locations (1):
- Applied Science Performance Institute, Tampa, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wright CJ, Arnold BL, Ross SE, Linens SW. Recalibration and validation of the Cumberland Ankle Instability Tool cutoff score for individuals with chronic ankle instability. Arch Phys Med Rehabil. 2014 Oct;95(10):1853-9. doi: 10.1016/j.apmr.2014.04.017. Epub 2014 May 9. PMID 24814563
- [Background] Ware J Jr, Kosinski M, Keller SD. A 12-Item Short-Form Health Survey: construction of scales and preliminary tests of reliability and validity. Med Care. 1996 Mar;34(3):220-33. doi: 10.1097/00005650-199603000-00003. PMID 8628042
- [Background] McKay AKA, Stellingwerff T, Smith ES, Martin DT, Mujika I, Goosey-Tolfrey VL, Sheppard J, Burke LM. Defining Training and Performance Caliber: A Participant Classification Framework. Int J Sports Physiol Perform. 2022 Feb 1;17(2):317-331. doi: 10.1123/ijspp.2021-0451. Epub 2022 Dec 29. PMID 34965513
- [Background] Balsalobre-Fernandez C, Varela-Olalla D. The Validity and Reliability of the My Jump Lab App for the Measurement of Vertical Jump Performance Using Artificial Intelligence. Sensors (Basel). 2024 Dec 10;24(24):7897. doi: 10.3390/s24247897. PMID 39771636